CLINICAL TRIAL: NCT06030791
Title: The Impact of Bone-tendon-bone Graft Harvest and Biological Regeneration of Bone-tendon Defects on the Development of Donor Site Morbidity After Anterior Cruciate Ligament Reconstruction
Brief Title: BTB Graft Harvest and Donor Site Morbidity After ACL Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Center of Vojvodina (Other)
Responsible Party: Principal Investigator, Mirko Obradovic, MD, Clinical Center of Vojvodina
Other Study IDs: MM12070106
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Anterior Cruciate Ligament Rupture; Donor Site Complication
Keywords: Anterior Cruciate Ligament Rupture; Autografts; Athletic Injuries; Magnetic Resonance Imaging
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: All examinees will undergo ACL reconstruction using BTB graft. MRI scans of operated knee will be conducted at two time points: 4 weeks and 1 year after ACL reconstruction surgery.
  Interventions: Diagnostic Test: MRI
- Group 2: All examinees will undergo ACL reconstruction using BTB graft. MRI scans of operated knee will be conducted at two time points: 4 weeks and 1 year after ACL reconstruction surgery.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI of operated knee

SUMMARY:
The aim of this observational study is to examine the connection between bone-tendinous defects after BTB graft harvest and the development of anterior knee pain.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the impact of bone-tendinous defects after ACL reconstruction on the development of anterior knee pain. We will assess the presence and extent of bone-tendinous defects using MRI scans, which will be conducted at two time points: 4 weeks and 1 year after ACL reconstruction surgery. Furthermore, we will compare the healing progress of the bone-tendinous defects observed on the MRI scans.

In addition, we will evaluate the correlation between the residual bone-tendinous defect and knee functionality by comparing the results with knee functional test (IKDC form, Lysholm score, Donor site morbidity score).

All individuals participating in the study have provided their informed consent by signing the necessary documents prior to their inclusion in the research.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients
* Diagnosed with ACL rupture based on medical history and clinical examination
* Confirmed ACL rupture on MRI scans
* A sufficient level of education to understand study procedures and be able to communicate with site personnel

Exclusion Criteria:

* Multiligament knee injuries
* Both knees injuries
* ACL re-rupture
* Postoperative complications in the form of infection

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: The study population will consist of individuals who have undergone ACL reconstruction surgery due to ligament injury. Participants will be recruited from the orthopedic clinic at University Clinical Center of Vojvodina. The inclusion criteria for this study are individuals aged 18 to 45 years old. Participants' medical records, including preoperative evaluations and surgical reports, will be reviewed to confirm eligibility and collect relevant baseline data.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Healing of bone-tendinous defect | 4 weeks postoperatively and 12 months postoperatively
  The healing progress will be assessed through MRI scans conducted at two time points: 4 weeks and 1 year after the surgical intervention. The measurement of bone-tendinous defect healing will be expressed both in cubic millimeters and as a percentage. The cubic millimeter measurement will quantify the size of the defect observed on the MRI scans. This measurement provides a precise assessment of the volume of the defect, allowing for accurate tracking of the healing process over time. In addition, the healing progress will also be expressed as a percentage, comparing the size of the defect at each time point relative to the initial defect size observed at the 4-week scan. This percentage calculation will offer a relative measure of the extent to which the bone-tendinous defect has healed or progressed over the course of the study.
Change of IKDC score | preoperatively and 12 months postoperatively
  The International Knee Documentation Committee (IKDC) form is a validated patient-reported outcome measure used to assess knee function and symptoms. It is a self-administered questionnaire that helps evaluate the subjective knee-related outcomes and overall knee function of individuals. The IKDC form covers various aspects, including symptoms, daily activities, sports and recreational activities, and knee-related quality of life. It consists of items that assess pain, stability, swelling, locking, giving way, range of motion, and the ability to perform specific tasks. Possible IKDC form score range from 0 to 100 and scores are divided into categories and interpreted based on cutoff values. Scores above 90 or 95 may be considered excellent or near-normal, scores between 80 and 89 may be considered good or satisfactory, scores between 70 and 79 may be considered fair or moderate, and scores below 70 may be considered poor or unsatisfactory.
Change of Lysholm score | preoperatively and 12 months postoperatively
  The Lysholm Knee Scoring Scale, often simply referred to as the Lysholm Score, is a patient-reported outcome measure used to evaluate the symptoms and functional limitations in individuals with knee injuries, especially those related to anterior cruciate ligament (ACL) damage. The Lysholm Score is commonly utilized in clinical practice and research to monitor the outcomes of knee surgeries or interventions. Categories Evaluated by Lysholm Knee Scoring Scale are: limping, using support, pain, locking, swelling, stair climbing, squatting and instability. The total score can range from 0 (severe symptoms and limitations) to 100 (no symptoms or limitations), with scores interpreted as Excellent, Good, Fair, or Poor based on the range they fall into.
Donor site morbidity score | 12 months postoperatively
  Donor site morbidity score is a new 10-question patient-oriented instrument that was developed to adequately assess morbidity at the site of BTB harvest. The intent was to measure subjective outcomes, including donor site pain, numbness, function, strength, and physical appearance at the surgical site. All questions had 4 possible answers, each representing increasing symptom severity and patient dissatisfaction. Answer choices were assigned 0 to 10 points depending on the severity or functional restriction. A perfect score of 100 represented no complaints whatsoever. Total scores were subdivided into 4 categories representing overall morbidity after surgery: excellent (≥93.3 points), good (80.0-93.2 points), fair (50.0-79.9 points), and poor (≤49.9 points).

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center of Vojvodina, Novi Sad, Serbia